CLINICAL TRIAL: NCT01695733
Title: Influenza Vaccination Response in Patients With Non-Hematological Malignancies
Brief Title: Response to Influenza Vaccine in Patients With Non-Hematologic Malignancies Receiving Chemotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no longer had funding to continue
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201010722
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Schedule A (Experimental): Influenza vaccination on the first day of chemotherapy
  Interventions: Biological: trivalent influenza vaccine
- Schedule B (Experimental): Influenza vaccination 1 week (+/- 1 day) prior to chemotherapy
  Interventions: Biological: trivalent influenza vaccine

INTERVENTIONS:
Biological: trivalent influenza vaccine
  Other Names: Flushield, Fluvirin, Fluzone, Influenza Vaccine

SUMMARY:
This clinical trial studies the best time to administer the influenza vaccine to patients with non-hematologic malignancies receiving chemotherapy. Giving the vaccine at different times relative to chemotherapy may affect how well it works to help the body build an immune response and prevent influenza in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have biopsy-confirmed non-hematological malignancy
* Patients must be scheduled to receive cytotoxic chemotherapy (adjuvant or metastatic setting), excluding immunotherapy
* Patients must be of age >=18 years.
* Patients must have an absolute lymphocyte count >= 1,000/mcL immediately prior to influenza vaccination
* Ability of the patient (or legally authorized representative if applicable) to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have already received the influenza vaccine during the season in which they are considered for eligibility will be excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the influenza vaccine or egg allergies
* Previous history of Guillian-Barre syndrome within the previous 6 weeks to influenza vaccination
* Patients must not be receiving chronic steroid therapy, defined as >= 14 days, unless used as part of a chemotherapy regimen
* Patients must not be on any other agents that can suppress the immune system
* Planned concurrent therapy with radiation
* Uncontrolled illness at time of enrollment or influenza vaccination including, but not limited to, ongoing or active febrile illness
* Psychiatric illness/social situations that would limit compliance with study requirements
* Known immunosuppression eg. history of organ transplantation or known human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because they may not be able to mount an appropriate immune response
* History of influenza-like illness, defined as a temperature > 37.8 degree C with cough or sore throat starting October 1, 2011 throughout the duration of the study
* Patient may not be scheduled to receive chemotherapy on a weekly basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Optimal timing of seasonal influenza vaccination with regard to chemotherapy administration schedule. | 4 weeks from the influenza vaccine
  We will assess co-primary endpoints of serologic response to the H3N2 and H1N1 strains in the 2011-2012 and 2012-2013 seasonal influenza vaccine.

SECONDARY OUTCOMES:
Report the presence of post-vaccination adverse events | 4 weeks from the influenza vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Saiama Waqar, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu